CLINICAL TRIAL: NCT02192372
Title: Impact of Metabolic Syndrome on Development of Contrast Induced Nephropathy After Elective Percutaneous Coronary Intervention
Brief Title: Metabolic Syndrome and Contrast Induced Nephropathy
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Özgür Ulaş Özcan, MD, Ankara University
Other Study IDs: MetS CIN
Record Dates: First submitted 2014-07-15; First posted 2014-07-16 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Contrast Induced Nephropathy; Metabolic Syndrome
Keywords: creatinine; glomerular filtration rate; metabolic syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- metabolic syndrome: Presence of 3 or more of these components: high fasting glucose (fasting serum glucose ≥ 100 mg/dl or drug treatment for elevated blood glucose), abdominal obesity (given as waist circumference > 102 cm in men and > 88 cm in women), high blood pressure (≥130/≥85 mmHg or drug treatment for hypertension), hypertriglyceridemia (serum triglycerides ≥150 mg/dl), low high-density lipoprotein cholesterol (<40 mg/dl in men and <50 mg/dl in women).
- control: Age and sex adjusted control subjects

SUMMARY:
Prevention of contrast induced nephropathy after interventional cardiologic procedures deserves close interest because of its association with prolonged hospitalization, increased cost and increased in hospital and long term mortality rates. An observational prospective cohort study was designed to determine whether metabolic syndrome predicts the development of contrast induced nephropathy after elective percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

Patients must be scheduled for elective percutaneous coronary intervention Clinical diagnosis of metabolic syndrome Patients must give informed consent

Exclusion Criteria:

Acute coronary events Acute renal failure End stage renal failure requiring hemodialysis Contrast allergy and exposure to nephrotoxic agent within 1 week before percutaneous coronary intervention Exposure to contrast agent within 1 week before the procedure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective percutaneous coronary intervention Patients with metabolic syndrome
Sampling Method: Non-Probability Sample
Enrollment: 599 (Actual)
Dates: Start 2014-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Contrast induced nephropathy | 24-48 hours after the percutaneous coronary intervention
  Contrast induced nephropathy was defined as an increase in serum creatinine of >25% or >0.5 mg/dl above the baseline value 24 or 48 hours after angiography.

SECONDARY OUTCOMES:
glomerular filtration rate | 48 hours after the percutaneous coronary intervention
  Glomerular filtration rate was estimated using the Cockcroft-Gault formula: (140-age) x weight (kg)/ serum creatinine (mg/dl) x 72 (x 0.85 for females)

OTHER OUTCOMES:
Cut-off point for baseline glomerular filtration rate to predict development of contrast induced nephropathy | baseline glomerular filtration rate

CONTACTS AND LOCATIONS:
Overall Officials: Ozgur Ulas Ozcan, Principal Investigator — Ankara University
Locations (1):
- Ankara University School Of Medicine, Department of Cardiology, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Ozcan OU, Adanir Er H, Gulec S, Ustun EE, Gerede DM, Goksuluk H, Tulunay Kaya C, Erol C. Impact of metabolic syndrome on development of contrast-induced nephropathy after elective percutaneous coronary intervention among nondiabetic patients. Clin Cardiol. 2015 Mar;38(3):150-6. doi: 10.1002/clc.22364. PMID 25800136